CLINICAL TRIAL: NCT05381688
Title: Respiratory Modulation by VIM Deep Brain Stimulation: N-of-1 Trial of Breath-holding and Peak Expiratory Flow
Brief Title: VIM DBS Respiratory Modulation: N-of-1 Trial
Status: Withdrawn | Type: Observational
Why Stopped: Covid prevented us from performing the study and the funding ran out
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: 256285/1
Record Dates: First submitted 2021-04-27; First posted 2022-05-19 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2022-05

CONDITIONS: Essential Tremor; Dystonic Tremor
MeSH Terms: conditions — Essential Tremor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ET VIM DBS patients: Essential tremor patients scheduled for VIM DBS
  Interventions: Procedure: VIM DBS
- DT VIM DBS patients: Dystonic tremor patients scheduled for VIM DBS
  Interventions: Procedure: VIM DBS

INTERVENTIONS:
Procedure: VIM DBS — Stereotactic deep brain stimulation of ventral intermediate nucleus of thalamus

SUMMARY:
Research from our group has demonstrated modulation of PEFR in patients with STN and PAG stimulation. However, the effect of VIM (motor thalamus) stimulation remains to be investigated. Our group has also been involved in research that indicates that VIM stimulation may reduce perception of breathlessness. However, methodological factors limit the conclusions that can be drawn from this prior work. N-of-1 trials, organised as a randomised multiphase crossover design, are uniquely well suited for DBS research where stimulation can be switched ON and OFF, and with simple tests that can be done quickly, multiple times. PEFR and breath-holding are simple tests that we will test in this way. Other respiratory tests will be carried out along side, as optional, in a single phase design. We aim to offer this study to a continuous cohort of patients scheduled to undergo VIM (ET/DT) DBS at our institution. We will establish a pre-operative baseline of respiratory function, and then perform the n-of-1 trial post-operatively, soon after the patient returns to hospital to receive their DBS programming.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for VIM DBS
* Diagnosis of ET or DT

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sequential cohort of patients with movement disorders (ET and DT) who are scheduled for VIM DBS at John Radcliffe Hospital. All will be contacted by a member of clinical care team for the study to be offered.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-09-09 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Breath-hold (urge to breath) | 3 months post-operative, ON and OFF: randomised, cross over, 5-phase design
  Time from start of breath-hold to urge to breathe

SECONDARY OUTCOMES:
Breath-hold (break point) | 3 months post-operative, ON and OFF: randomised, cross over, 5-phase design
  Time from start of breath-hold to breakpoint
Peak Expiratory Flow Rate | 3 months post-operative, ON and OFF: randomised, cross over, 5-phase design
  Maximum PEFR of three trials
Dyspnoea-12 Questionnaire | Baseline and 3 months post-operative
  Difference in D12 score
Oscillometry | Baseline and 3 months post-operative ON and OFF
  Difference in airway resistance
Maximum inspiratory pressure | Baseline and 3 months post-operative ON and OFF
  Best MIP of three trials

CONTACTS AND LOCATIONS:
Overall Officials: Alex L Green, FRCS, Principal Investigator — University of Oxford

IPD SHARING:
Plan to Share IPD: Undecided